CLINICAL TRIAL: NCT06751316
Title: Clinical and Radiographic Evaluation of MTA Pulpotomy Versus Conventional Pulpectomy in Primary Molars With Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of MTA Pulpotomy Versus Conventional Pulpectomy in Primary Molars With Irreversible Pulpitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeyad Nasr Abdelhafeiz, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pulpotomy Versus Pulpectomy
Record Dates: First submitted 2024-12-10; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Decayed Primary Molars With Irreversible Pulpitis
Keywords: MTA pulpotomy; Pulpectomy; Decayed primary molars; Irreversible pulpitits

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Pulpectomy (Experimental): Conventional pulpectomy using Zinc Oxide/Eugenol
  Interventions: Procedure: Conventional Pulpectomy
- MTA Pulpotomy (Experimental): Pulpotomy using MTA
  Interventions: Procedure: MTA Pulpotomy

INTERVENTIONS:
Procedure: Conventional Pulpectomy — Removal of radicular pulp tissue, placing Zinc Oxide/Eugenol and covered by stainless steel crown
  Arms: Conventional Pulpectomy
Procedure: MTA Pulpotomy — Removal of coronal pulp tissue, placing MTA and covered by stainless steel crown
  Arms: MTA Pulpotomy

SUMMARY:
This study is designed to compare between MTA Pulpotomy (Removal of coronal pulp tissue, placing MTA and covering with Stainless steel crown) Versus Conventional Pulpectomy (Removal of radicular pulp tissue, placing Zinc Oxide/Eugenol and covering with Stainless steel crown) in irreversible pulpitis in primary second molars.

ELIGIBILITY:
Inclusion Criteria:

* Patients:
* Aged 4-7 years, cooperative, in good general health and medically within normal
* Teeth:
* Restorable mandibular second primary molars.
* History of irreversible pulpitis.
* Preoperative radiograph:
* Absence of periapical or inter-radicular radiolucency.
* Absence of widening of periodontal ligaments (PDL) space.
* Absence of internal or external root resorption.

Exclusion Criteria:

* Patients:
* With systemic disorders.
* Physical or mental disabilities.
* Unable to attend follow- up visits.
* Refusal of Participation.
* Refusal to sign the informed consent.
* Teeth:
* Previously accessed teeth.
* Mobile mandibular second primary molar.
* Swelling in the vestibule or on palpation.
* Pain on percussion.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
• rate of clinical success | 12 months
  * tenderness on percussion and palpation
  * sinus/parulis/fistula
  * soft tissue swelling
  * pathological mobility

SECONDARY OUTCOMES:
• rate of radiographic success | 12 months
  * pathologic root resorption.
  * interradicular and/or periapical radiolucency

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR